CLINICAL TRIAL: NCT04042428
Title: Generation of Biological Samples Positive to Somatropin for Anti-doping Control
Acronym: GH5
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IMIMFTCL/GH/5
Record Dates: First submitted 2019-07-31; First posted 2019-08-02 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2019-07

CONDITIONS: Healthy Volunteers
Keywords: Somatropin; Growth hormone; Anti-doping control; Athletic performance
MeSH Terms: interventions — Human Growth Hormone

STUDY DESIGN:
Intervention Model Description: Samples from treatment group are compared to samples from control group (not receiving treatment). It is not possible to use a basal sample of the subjects receiving treatment as a comparator since a minimum period of 2 months' time is required between a 450 mL extraction and another.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Subjects receive a 14-day treatment. A 450 mL blood sample is extracted 6 hours after the last administration (day 14).
  Interventions: Drug: Somatropin injection
- Control group (No Intervention): Subjects do not receive any treatment. A 450 mL blood sample is extracted at baseline.

INTERVENTIONS:
Drug: Somatropin injection — Subjects receive a daily subcutaneous dose of 0.2 IU/kg (0.067 mg/kg) of recombinant somatropin (rhGH) during 14 days.
  Arms: Treatment group

SUMMARY:
Background:

Somatropin, also known as recombinant growth hormone (rhGH), is one of the World Anti-Doping Agency (WADA) prohibited substances. Its consumption in athletes has been banned since 1990, as it is known to improve physical performance.

Hypothesis:

The subcutaneous administration of recombinant somatropin (rhGH) in healthy subjects allows obtaining positive doping samples.

The concentrations of hGH variants (isoforms) and biomarkers can be measured in serum.

Objectives:

Primary objective: To generate enough serum samples positive to recombinant somatropin in order to be analyzed as control samples by anti-doping laboratories.

Secondary objective: To determine the analytical parameters necessary to detect the administration of recombinant somatropin in healthy volunteers by direct and/or indirect methods.

Methods:

Phase I, open, randomized clinical trial, with a treatment condition (recombinant somatropin or rhGH) administered subcutaneously to 4 subjects (2:1 ratio). Control samples of the study correspond to basal samples of 2 subjects who do not receive any treatment.

DETAILED DESCRIPTION:
A blood sample volume of 450 mL is obtained from each subject receiving the treatment condition to perform the proposed tests.

In order to validate the determination methodology of hGH variants and biomarkers, blood samples from treatment group subjects are compared to reference blood samples of 450 mL from a control group (not receiving treatment) as it is not possible to obtain a basal sample of such volume from the subjects receiving treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male volunteers between 20 and 30 years old.
* History and physical examination that demonstrate not presenting organic or psychiatric disorders.
* ECG, blood and urine tests performed before the trial within normal limits. Minor or punctual variations of these limits will be allowed if, in the opinion of the principal investigator, they have no clinical significance, do not pose a risk to the subject and do not interfere in the evaluation of the product. These variations and their non-relevance will be justified in writing.
* Body mass index [BMI: weight/height^2] between 19 and 26, and weight between 50 and 90 kg.
* Able to understand and accept the trial procedures and sign an informed consent.

Exclusion Criteria:

* Failure to meet the inclusion criteria.
* Having suffered some organic disease or major surgery during the three months prior to the trial.
* Suffering any type of illness, acute or chronic at the time of the study.
* Background or clinical evidence of cardiovascular, respiratory, renal, hepatic, endocrine, gastrointestinal, hematological, neurological, dermatological, or other acute or chronic diseases that, in the opinion of the Principal Investigator or the collaborators designated by it, may pose a risk for the subjects, may interfere with the objectives of the study, or may suggest an alteration in the absorption, distribution, metabolism or excretion of the drug.
* Having suffered some kind of bone or ligament injury in the last three years.
* History or clinical evidence of psychiatric disorders, alcoholism, drug abuse or addiction to other substances (except for nicotine) or regular consumption of psychoactive drugs. With regard to nicotine, consumers of more than 10 cigarettes/day will be excluded.
* Alcohol consumption over 15 g/day in men and 10 g/day in women.
* Consumers of more than 3 cups of coffee and/or tea per day, consumers of more than 3 units of cola, other stimulant drinks or equivalent per day, in the 2 months prior to the start of the study.
* Regular intake of medication in the month preceding the study. Other kinds of medication may be admitted at the discretion of the Investigator.
* Having donated blood or participated in studies in which there were blood draws in the previous 4 weeks.
* History of allergy, idiosyncrasy, hypersensitivity or adverse reactions to the active principle or any of the excipients. Serious adverse drug reactions.
* Having participated in another clinical trial with medication in the three months prior to the start of the study.
* Subjects with contraindications to treatment with the study drug (according to the summary of product characteristics).
* Positive serology to hepatitis B, C or HIV.
* Being unable to understand the nature, consequences of the trial and the procedures that are asked to follow.

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2019-10-25 (Actual); Primary Completion 2020-01-08 (Actual); Study Completion 2020-01-08 (Actual)

PRIMARY OUTCOMES:
Seric concentration of rhGH | 6 hours after last administration
  Concentration of the pool of molecular variants (isoforms) of somatropin in blood

SECONDARY OUTCOMES:
Changes in the proportion of somatropin isoforms | 6 hours after last administration
  Variation of the concentration in blood of each somatropin isoform after rhGH administration
Changes in seric concentration of ghrelin | 6 hours after last administration
  Variation of seric concentration of ghrelin (biomarker) in blood after rhGH administration
Changes in seric concentration of leptin | 6 hours after last administration
  Variation of seric concentration of leptin (biomarker) in blood after rhGH administration
Changes in seric concentration of adiponectin | 6 hours after last administration
  Variation of seric concentration of adiponectin (biomarker) in blood after rhGH administration
Changes in seric concentration of type III procollagen (P-III-P) | 6 hours after last administration
  Variation of seric concentration of type III procollagen (biomarker) in blood after rhGH administration
Changes in seric concentration of cross-linked C-terminal telopeptide of type I collagen (ICTP) | 6 hours after last administration
  Variation of seric concentration of cross-linked C-terminal telopeptide of type I collagen (biomarker) in blood after rhGH administration
Changes in seric concentration of Insulin-like Growth Factor I (IGF-I) | 6 hours after last administration
  Variation of seric concentration of Insulin-like Growth Factor I (biomarker) in blood after rhGH administration
Changes in seric concentration of Insulin-like Growth Factor Binding Protein 3 (IGFBP-3) | 6 hours after last administration
  Variation of seric concentration of Insulin-like Growth Factor Binding Protein 3 (biomarker) in blood after rhGH administration

CONTACTS AND LOCATIONS:
Overall Officials: Ana M Aldea Perona, Dr, Principal Investigator — IMIM (Hospital del Mar Medical Research Institute)
Locations (1):
- IMIM (Hospital del Mar Medical Research Institute), Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No